CLINICAL TRIAL: NCT01582347
Title: A Randomized, Double-blind, Double-dummy, Active-drug-controlled, Parallel-group, Multicentre Acceptability and Safety Study of the Transfer From Subutex/Suboxone to RBP-6300 in Opioid-dependent Subjects
Brief Title: Transfer of Subjects From Subutex/Suboxone to RBP-6300
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RB-UK-11-0017
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Opioid Related Disorder
Keywords: Opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naloxone; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RBP-6300 (Experimental): During the Double-Blind Transfer Period (Days 1-7), participants take RBP-6300 at a level (either 10, 20 or 30 mg/day) equivalent to dosing during the Run-In Period, plus Placebo for Subutex®/Suboxone®. This is followed by a 3-day Transition Period (Days 8-10) in which participants take active Subutex®/Suboxone® equal to the dose taken during the Run-In Period plus placebo matching RBP-6000.
  Interventions: Drug: RBP-6300; Drug: Subutex®/Suboxone®; Drug: Placebo for RBP-6300; Drug: Placebo for Subutex®/Suboxone®
- Subutex®/Suboxone® (Active Comparator): During the Double-Blind Transfer Period (Days 1-7), participants take Subutex®/Suboxone® at a level (either 8, 16 or 240 mg/day) equivalent to dosing during the Run-In Period, plus Placebo for RBP-6000. This is followed by a 3-day Transition Period (Days 8-10) in which participants take active Subutex®/Suboxone® equal to the dose taken during the Run-In Period plus placebo matching RBP-6000.
  Interventions: Drug: Subutex®/Suboxone®; Drug: Placebo for RBP-6300

INTERVENTIONS:
Drug: RBP-6300 — Participants randomized to the RBP-6300 treatment arm take either 10, 20 or 30 mg/day RBP-6300 tablets during the Transfer Period (study days 1-7).
  Oral RBP-6300 tablets containing 10 mg buprenorphine hemiadipate HCl and 10 mg naloxone HCl dehydrate.
  Other Names: buprenorphine hemiadipate HCl; naloxone HCl
  Arms: RBP-6300
Drug: Subutex®/Suboxone® — Participants randomized to the Subutex®/Suboxone® treatment arm take the dosage of either drug on which they were previously stabilised during the Run-In, Transfer, and Transition Periods.
  Participants randomized to the RBP-6300 treatment arm take the dosage of either drug on which they were previously stabilised during the Run-In and Transition Periods.
  Sublingual Subutex® tablets containing 8 mg buprenorphine and and sublingual Suboxone® tablets containing 8 mg buprenorphine and 2 mg naloxone.
  Other Names: buprenorphine; naloxone
Drug: Placebo for RBP-6300 — Participants randomized to the Subutex®/Suboxone® treatment arm take Placebo for RBP-6300 during the Transfer and Transition Periods.
  Participants randomized to the RBP-6300 treatment arm take Placebo for RBP-6300 during the Transition Period.
  Other Names: placebo
Drug: Placebo for Subutex®/Suboxone® — Participants randomized to the RBP-6300 treatment arm take Placebo for Subutex®/Suboxone® during the Transfer Period.
  Other Names: placebo
  Arms: RBP-6300

SUMMARY:
This study is designed to determine if opioid dependent subjects who are already receiving Subutex and/or Suboxone can transfer to RBP-6300. Upon completing the study, subjects will continue their pre-study prescribed dosage of Subutex and/or Suboxone

DETAILED DESCRIPTION:
During the open-label Run-In Period (study days -7 to -1), participants receive Subutex®/Suboxone® at one of three dose levels, depending on the dose level for that subject on entry to the study: 8 mg/day, 16 mg/day, or 24 mg/day.

During the 7-day, active drug-controlled, double-blind Transfer Period (study days 1-7), participants are randomized to either Subutex®/Suboxone® or RBP-6300 active drug at dosing levels equivalent to the level during the Run-In Period plus placebo matching the other drug.

This is followed by a 3-day single-blind Subutex®/Suboxone® Transition Period in which participants receive the same dose given during the Run-In Period.

ELIGIBILITY:
Inclusion Criteria:

* Be Male or non-pregnant, non-lactating females
* Be at least 18 years of age
* Meet Diagnostic and Statistical Manual of Mental Disorders, DSM-IV-TR (Diagnostic and Statistical Manual-IV-TEXT REVISION)criteria for opioid dependence at screening
* Be on stable dose of 8, 16, or 24mg/day for about 30 days prior to screening
* Female subjects of childbearing potential must have a negative urine test prior to enrollment into the study

Exclusion Criteria:

* Have participated in an experimental drug or device study within the last 60 days
* If female, be breast feeding or lactating
* Have any medical condition that in the opinion of the physician investigator would preclude the subject from completing the study
* Have a clinically significant abnormal finding (in the opinion of the investigator)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Treatment | 7 days
  To demonstrate that RBP-6300 is not inferior to Subutex/Suboxone as assessed by the peak change from baseline in the pre-dose COWS score during the double-blind transfer phase

SECONDARY OUTCOMES:
Assess the overall clinical response to RBP-6300 | one year
  One of the secondary objectives is to evaluate the safety and tolerability of RBP-6300 in terms of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Scherbaum, Prof. Dr., Principal Investigator — Medical University, Duisburg-Essen, Germany; Michael Wolzt, Prof. Dr., Principal Investigator — Univ.-Klinik fur Klinische Pharmakologie, AKH Wien, Wien; Wolfgang Fleischhacker, Prof. Dr., Principal Investigator — Medical University Innsbruck; Vratislav Rehak, Dr., Principal Investigator — Remedis s.r.o., Prague; Zdenka Stankova, Dr., Principal Investigator — Masaryk Hospital Usti nad Labem; Oliver Pogarell, PD. Dr., Principal Investigator — Medical University, Munich; Bernd Weber, Dr., Principal Investigator — Praxis Dr. Bernd Weber am Koenigsplatz Schwerpunkprax is fur Suchtmedizin, Kassel; Edith Issler, Dr., Principal Investigator — Infectomed GbR Zentrum fuer medizinische Studien, Stuttgart; Wieland Tietje, Dr., Principal Investigator — Drs. Tieje, Heer & Koc, Bremen; Eduard Boniakowski, Dr., Principal Investigator — Psychosoziale Begleitung - Praxis Boniakowski, Regensburg; Charlotte Rechenmacher, Dr, Principal Investigator — Praxis Dr. Rechenmacher, Oldenburg; Georgieva, Dr., Principal Investigator — Karolinska Institute, Stockholm; Spyridon Kilaidakis, Dr., Principal Investigator — Region Örebro County; Claus Schubert, Dr, Principal Investigator — Substitutionsambulanz Geinhausen; Chaim Jellinek, Principal Investigator — a.i.d., Ambulanz fur integrierte Drogenhilfe; Karl Heinz Meller, Dr, Principal Investigator — Praxis Dr. Meller
Locations (15):
- Austria (4):
  - Prof. Dr. Fleischhacker, Austria
  - Dr. Lindenbauer, Linz
  - Prof. Dr. Wurst, Salzburg
  - Prof. Wolzt, Vienna
- Czechia (2):
  - Dr. Vehak, Prague
  - Dr. Stankova, Ústí nad Labem
- Germany (7):
  - Dr. Tietje, Bremen
  - Prof. Scherbaum, Essen
  - Dr. Weber, Kassel
  - PD. Dr. Pogarell, Munich
  - Dr. Rechenmacher, Oldenburg
  - Dr. Boniakowski, Regensburg
  - Dr. Issler, Stuttgart
- Sweden (2):
  - Dr. Kilaidakis, Örebro
  - Dr. Georgieva, Stockholm